NCT05430022 GROUP DEPRESSION TREATMENT FOR AUTISTIC YOUTH July 14, 2022

## ADAPTED COGNITIVE BEHAVIORAL THERAPY FOR DEPRESSION IN YOUTH WITH AUTISM

## STATISTICAL ANALYSIS PLAN

- Feasibility: Attrition proportion (i.e., frequencies) of youth who complete the study and proportion of youth who withdraw from study and reasons listed.
- Preliminary Efficacy: One-way ANOVAS and/or linear mixed models will be used to assess
  change in adolescent depressive symptom severity on the Revised Children's Anxiety and
  Depression Scale (RCADS), self- and parent-report versions. Potential changes in depressive
  symptom severity may provide preliminary support of the potential efficacy of the intervention.